CLINICAL TRIAL: NCT02596256
Title: Apatinib Plus Docetaxel Versus Docetaxel as Second-line Treatment in Advanced Gastric Cancer Stage II Randomized Controlled Clinical Studies
Brief Title: Apatinib Plus Docetaxel Versus Docetaxel as Second-line Treatment in Advanced Gastric Cancer (AHEAD-301)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Guanghai, Department Director, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-301
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Experimental): Apatinib Mesylate Tablets (500 mg qd p.o.) and Docetaxel (60mg/m2 i.v. d1 q21d)
  Interventions: Drug: Apatinib; Drug: Docetaxel
- contrast group (Active Comparator): Docetaxel (60mg/m2, i.v. d1 q21d)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Apatinib — Apatinib (500 mg qd p.o.) until disease progression or intolerable toxicity
  Other Names: ATAN
  Arms: control group
Drug: Docetaxel — Docetaxel (60 mg/m2 qd d1 q3w i.v.) until disease progression or intolerable toxicity

SUMMARY:
Apatinib plus docetaxel versus docetaxel as second-line treatment in advanced gastric cancer.

DETAILED DESCRIPTION:
This trial investigated the safety and efficacy of apatinib plus docetaxel, as a treatment option for heavily pretreated patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: more than 18 years old, male or female;
2. Pathologically diagnosed with advanced gastric cancer (including adenocarcinoma of the gastroesophageal junction) with measurable metastases outside the stomach (measuring ≥ 10mm on spiral computed tomography(CT) scan, satisfying the criteria in Response Evaluation Criteria In Solid Tumors (RECIST) 1.1);
3. Failure of prior therapy (during or after treatment) in patients who have received at first line chemotherapy regimens(platinum - based regimens);
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1;
5. Major organ function has to meet the following criteria; (1) For results of blood routine test and biochemical tests:

   1. Hemoglobin (HB) ≥ 80g / L,
   2. ANC ≥ 1.5 × 109 / L,
   3. PLT ≥ 90 × 109 / L,
   4. ALT and AST ≤ 2.5 × ULN, liver metastases, if any, the ALT and AST≤5 × ULN,
   5. Bilirubin ≤ 1.5 times the upper limit of normal (ULN),
   6. Serum creatinine ≤ 1.5 times the upper limit of normal (ULN),
   7. Serum albumin ≥ 30g / L;
6. An expected survival of ≥ 3 months;
7. Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative. They shall take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men, (previous surgical sterilization accepted), shall agree to take appropriate methods of contraception during the study until the 8th week post the last administration of study drug;
8. Patient has to voluntarily join the study and sign the Informed Consent Form for the study.

Exclusion Criteria:

1. Confirmed that apatinib and/or its accessories allergy;
2. Subjects with poor-controlled arterial hypertension (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg) despite standard medical management; Coronary heart disease greater than Class Ⅰ; Ⅰ-level arrhythmia (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms) together with Class Ⅰ cardiac dysfunction; Patients with positive urinary protein;
3. Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
4. Subjects with high gastrointestinal bleeding risk, including the following conditions: local active ulcer lesions with positive fecal occult blood test (++); history of black stool, or vomiting blood in the past 2 months;unresected primary lesion in stomach with positive fecal occult blood test (+), ulcerated gastric carcinoma with massive alimentary tract bleeding risk judged by PIs based on gastric endoscopy result;
5. Abnormal Coagulation (INR>1.5、APTT>1.5 UNL), with tendency of bleed;
6. Associated with CNS (central nervous system) metastases;
7. Pregnant or lactating women;
8. Pts with other malignant tumor within 5 years;
9. With psychotropic drug abuse history and can't get rid of or mental disorder patients;
10. Participated in other clinical trials within 4 weeks;
11. Pts received VEGFR inhibitor treatment(i.e. sorafenib, sunitinib);
12. Any other condition that might place the patient at undue risk or preclude a patient from completing the study;
13. Other conditions regimented at investigators' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China